CLINICAL TRIAL: NCT02560350
Title: Implantation of a Small Intestinal Submucosa Scaffold Combined With Adipose-derived Stem Cells to Evaluate Its Potential to Form an Adipocyte-containing Hypodermis
Brief Title: Small Intestinal Submucosa Scaffold Combined With Adipose-derived Stem Cells to Form an Adipocyte-containing Hypodermis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2015-090
Record Dates: First submitted 2015-09-01; First posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Adipogenesis
Keywords: adipose-derived stem cells; small intestinal submucosa; adipocyte-containing hypodermis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Human adipose tissues were obtained from five healthy adult women who underwent abdominal liposuction. They were aged 28 to 45 years (mean, 32.15±4.8 years) and had no infectious or endocrine diseases. Ten millilitres of discarded adipose tissue from the humans was used to gain the adipose-derived stem cells. In this study, the investigators will evaluate the potential of a small intestinal submucosa scaffold combined with adipose-derived stem cells to form an adipocyte-containing hypodermis.

DETAILED DESCRIPTION:
Human adipose tissues were obtained from five healthy adult women who underwent abdominal liposuction. They were aged 28 to 45 years (mean, 32.15±4.8 years) and had no infectious or endocrine diseases. All protocols using human samples were approval by the Institutional Review Board of Nanfang Hospital (no.18502), and samples were obtained with written informed consent. Ten millilitres of discarded adipose tissue from the humans was washed extensively with equal volumes of phosphate-buffered saline (PBS); minced into a fine, homogeneous preparation; and digested at 37°C for 30 min with 0.125% type I collagenase. Enzyme activity was neutralized with Dulbecco's modified Eagle's medium (DMEM) containing 10% FBS. Then, the sample was filtered through a 200-mm nylon mesh to remove cellular debris and was centrifuged at 1500 revolutions per minute (rpm) for 5 min. The precipitate was resuspended in 6~10 ml NH4Cl and incubated at room temperature for 10 min to lyse contaminating red blood cells. The compound was centrifuged at 1500 rpm for an additional 5 min. The ASCs were collected via centrifugation as described above, resuspended in 2 ml of control medium (DMEM containing 10% FBS and 1% antibiotic/antimycotic solution) and incubated at 37°C in a humidified chamber containing 5% CO2 for 48 h. Next, the plates were washed extensively with PBS to remove residual non-adherent red blood cells and debris. The resulting cell population was termed ASCs, and the cultures were expanded with media changes at 3-day intervals. Cells at passage 1 through 6 were used for all experiments.

ELIGIBILITY:
Inclusion Criteria:

* healthy people with no infectious diseases
* healthy people with no endocrine diseases

Exclusion Criteria:

* sick people

Ages: 28 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy people with normal adipose tissue
Sampling Method: Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The adipogenesis of adipose-derived stem cells combined with the small intestinal submucosa by histological observation | up to 12 months
  From 2015-9 to 2016-9

SECONDARY OUTCOMES:
The proliferation of adipose-derived stem cells after seeding on the SIS scaffold by MTT method | up to 12 months
  From 2015-9 to 2016-9
The adhesion of adipose-derived stem cells after seeding on the SIS scaffold by histological observation | up to 12 months
  From 2015-9 to 2016-9

CONTACTS AND LOCATIONS:
Overall Officials: Ping Jiang, PhD, Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China